CLINICAL TRIAL: NCT03104335
Title: Apatinib for Advanced Soft Tissue Sarcoma Patients After Failure of Traditional Therapy: an One-armed, Phase 2, Open-label, Multicenter Prospective Trial
Brief Title: Apatinib for Advanced Soft Tissue Sarcoma Patients: a Phase 2, Multicenter Trial
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Not enough patients
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking University Shougang Hospital (Other); Peking University International Hospital (Other)
Responsible Party: Principal Investigator, GUO WEI, Director of Musculoskeletal Tumor Center and Principal Investigator of this study, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PekingUAH-sarcoma070330
Record Dates: First submitted 2017-04-02; First posted 2017-04-07 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Soft Tissue Sarcoma Adult; Advanced Cancer
Keywords: soft tissue sarcoma; advanced; apatinib; tyrosine-kinase inhibitors
MeSH Terms: conditions — Sarcoma | interventions — apatinib

STUDY DESIGN:
Intervention Model Description: participants will be advised to recieve 750 mg daily once apatinib for body surface area (BSA) > 1.5 and 500mg daily for BSA <1.5. Half an hour after meal and everyday at the same time is usually advised.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm (Experimental): every participant will recieve 750 mg daily once oral administration of apatinib for body surface area (BSA) > 1.5 and 500mg daily for BSA <1.5. Half an hour after meal and everyday at the same time is usually advised.
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — 750 mg daily once oral administration of apatinib for body surface area (BSA) > 1.5 and 500mg daily for BSA <1.5. Half an hour after meal and everyday at the same time is usually advised.
  Other Names: apatinib mesylate tablets

SUMMARY:
Patients with advanced soft tissue sarcoma(rhabdomyosarcoma and liposarcoma excluded), who experience progression after standard chemotherapy, have limited treatment options which promise a survival benefit.This trial tends to explore apatinib, which is a domestic highly selective inhibitor of vascular endothelial growth factor receptor-2, as a treatment option for heavily pretreated soft tissue sarcoma patients.

DETAILED DESCRIPTION:
From April 1st 2017 to June 1st 2019, participants who met the following criteria were included: 1) histologically confirmed high-grade soft tissue sarcoma(rhabdomyosarcoma and liposarcoma excluded); 2) initial treated in the orthopedic oncology departments of three affiliated hospitals of Peking University,including Peking University People's Hospital, Peking University Shougang Hospital and Peking University International Hospital; 3) not amenable to curative treatment; 4) multiple metastatic lesions which could not be cured by local therapy or unresectable local advanced lesions; 5) having measurable lesions according to Response Evaluation Criteria for Solid Tumors 1.1(RECIST 1.1); 6) expected to live longer than 3 months with an Eastern Cooperative Oncology Group performance status of 0 or 1 and acceptable hematologic, hepatic, and renal function; 7) needed to be verified refractory to doxorubicin and ifosfamide.

All those participants need to sign informed consent forms for data collection and use for research purpose before inclusion, of which children patients' informed forms should be signed by their legal parents. Once the patient registered, he/she will be evaluated by his/her doctors of these departments at the clinic, and his/her follow-up should be done every eight weeks with at least chest CT as well as imaging of tumor lesions at other sites. A follow-up file should be sent every eight weeks to the coordination desk of these departments. This study was approved by the institutional review board, Peking University People's Hospital, Peking University Shougang Hospital and Peking University International Hospital Ethics Committee for Clinical Investigation, and conducted in accordance with the Declaration of Helsinki and Good Clinical Practice.

The investigators demand patients to use at least doxorubicin and ifosfamide. In a phase I trial, apatinib (Jiangsu Hengrui Medicine, Lianyungang, China) showed good oral bioavailability at a dose of 850 mg a day, the maximum-tolerated dose. Considering this, the participants are designed to receive 750 mg daily once oral administration of apatinib for body surface area (BSA) > 1.5 and 500mg daily for BSA <1.5. If the investigators meet with treatment interruptions because of grade 3 hematologic or grade 2 non-hematologic toxicities, dose reductions to 750 mg or 500 mg of apatinib per day, and supportive care should be allowed for the management of adverse events (AEs).

The primary objective is to describe the efficacy of apatinib in sarcoma patients. Endpoints is objective response rate (CR+PR) and Progression-Free-Survival (PFS) for each protocol as described containing apatinib according to RECIST 1.1. The secondary objective is overall survival (OS), duration of response (DR) and the characterization of toxicities. PFS is defined as the time from the start of using apatinib until disease progression or death, whichever occurs first. OS is defined as the time from the start of using apatinib until death. The period from appearance of response or stable disease to progression or death is thus considered the duration of response (DR).

Safety evaluation will be based on the frequency and severity of toxicities graded according to the Common Terminology Criteria for Adverse Events.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically and/or cytologically confirmed soft tissue sarcoma(rhabdomyosarcoma and liposarcoma excluded) who are resistant / refractory to approved therapies or for whom no curative therapies are available.
* All previous treatment (including surgery, radiotherapy and systemic anti-neoplastic therapy) must have been completed at least three weeks prior to study entry and any acute toxicities must have resolved.
* Aged >/= 16 years.
* Eastern Cooperative Oncology Group (ECOG) performance status score of </= 2.
* Written informed consent prior to any study specific screening procedures with the understanding that the patient may withdraw consent at any time without prejudice.
* Willing and able to comply with the protocol guidelines for the duration of the study.

Exclusion Criteria:

* Unstable metastases to the central nervous system (CNS).
* tumor embolus located at pulmonary vein.
* Any of the following laboratory parameters: a) hemoglobin < 9 g/dL (5.6 mmol/L); b) neutrophils <1.5 x 109/L; c) platelets <100 x 109/L; d) serum bilirubin >25 µmol/L (1.5 mg/dL); e) liver function tests with values >3 x upper limit of normal (ULN) f) serum creatinine >1.5 x ULN or creatinine clearance < 60 mL/minute.
* Positive history of HIV, active hepatitis B or active hepatitis C or severe/uncontrolled intercurrent illness or infection
* Clinically significant cardiac impairment or unstable ischemic heart disease including a myocardial infarction within six months of study start
* Patients with marked Baseline prolongation of QT/QTc interval (QTc interval > 450 msec for males or > 470 msec for females) using the Fridericia method for QTc analysis
* Bleeding or thrombotic disorders, or using therapeutic dosages of anticoagulants, such as warfarin. Occasional use of NSAIDs and antiplatelet agents such as aspirin, clopidogrel, aggrenox and dipyridamole are not considered exclusionary only if INR>1.5 or prothrombin time（PT）>ULN+4s or activated partial thromboplastin time (APTT) >1.5 ULN.
* Requirement for chronic use of full dose aspirin or non-steroidal anti-inflammatory drugs (NSAIDs)
* Poorly controlled hypertension (defined as requiring changes in any hypertensive regimen within 1 week of study entry) or patients diagnosed with hypertension based on repeat blood pressure measurements of >160/90 mmHg at Screening
* Proteinuria > 1+ on urine dipstick testing or 30 mg/dL
* A history of gastrointestinal malabsorption or having undergone surgery requiring gastrointestinal anastomoses within four weeks of starting therapy or who have not recovered from major surgery within three weeks of starting therapy History of alcoholism, drug addiction, or any psychiatric or psychological condition which, in the opinion of the Investigator, would impair study compliance.
* Any treatment with investigational drugs within 30 days before the start of the study
* Previous treatment with apatinib or other anti-angiogenesis tyrosine kinase inhibitors
* receive CYP3A4 inhibitors within 7 days or CYP3A4 inducers within 12 days.
* uncontrollable complicated diseases: such as infectious diseases, diabetes mellitus and so on.
* Women who are pregnant or breast-feeding; women of childbearing potential with a positive pregnancy test at Screening or no pregnancy test. Women of childbearing potential unless (1) surgically sterile or (2) using adequate measures of contraception (including two forms of contraception, one of which must be a barrier method) in the opinion of the Investigator. Perimenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
* Fertile males with female partners who are not willing to use contraception or whose female partners are not using adequate contraceptive protection
* Legal incapacity

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 4 months
  the number of participats (complete response+ partial response according to RECIST 1.1)/ total participants number

SECONDARY OUTCOMES:
Duration of Response (DR) | 4 months and 6 months
  The period from appearance of response or stable disease to progression or death is thus considered the duration of response (DR).
Progression-Free Survival(PFS) | 6 months
  PFS is defined as the time from the start of using apatinib until disease progression or death, whichever occurred first.
Overall Survival(OS) | 12 months
  OS is defined as the time from the start of using apatinib until death

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, M.D.Ph.D., Principal Investigator — Musculoskeletal Tumor Center of Peking University People's Hospital
Locations (3):
- China (3):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - Peking University International Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jo VY, Doyle LA. Refinements in Sarcoma Classification in the Current 2013 World Health Organization Classification of Tumours of Soft Tissue and Bone. Surg Oncol Clin N Am. 2016 Oct;25(4):621-43. doi: 10.1016/j.soc.2016.05.001. Epub 2016 Jul 30. PMID 27591490
- [Background] Brodowicz T, Liegl-Atzwager B, Tresch E, Taieb S, Kramar A, Gruenwald V, Vanseymortier M, Clisant S, Blay JY, Le Cesne A, Penel N. Study protocol of REGOSARC trial: activity and safety of regorafenib in advanced soft tissue sarcoma: a multinational, randomized, placebo-controlled, phase II trial. BMC Cancer. 2015 Mar 14;15:127. doi: 10.1186/s12885-015-1143-y. PMID 25884155
- [Background] Bains R, Magdum A, Bhat W, Roy A, Platt A, Stanley P. Soft tissue sarcoma - A review of presentation, management and outcomes in 110 patients. Surgeon. 2016 Jun;14(3):129-35. doi: 10.1016/j.surge.2014.06.002. Epub 2014 Sep 30. PMID 25261278
- [Background] Sleijfer S, Ray-Coquard I, Papai Z, Le Cesne A, Scurr M, Schoffski P, Collin F, Pandite L, Marreaud S, De Brauwer A, van Glabbeke M, Verweij J, Blay JY. Pazopanib, a multikinase angiogenesis inhibitor, in patients with relapsed or refractory advanced soft tissue sarcoma: a phase II study from the European organisation for research and treatment of cancer-soft tissue and bone sarcoma group (EORTC study 62043). J Clin Oncol. 2009 Jul 1;27(19):3126-32. doi: 10.1200/JCO.2008.21.3223. Epub 2009 May 18. PMID 19451427
- [Background] van der Graaf WT, Blay JY, Chawla SP, Kim DW, Bui-Nguyen B, Casali PG, Schoffski P, Aglietta M, Staddon AP, Beppu Y, Le Cesne A, Gelderblom H, Judson IR, Araki N, Ouali M, Marreaud S, Hodge R, Dewji MR, Coens C, Demetri GD, Fletcher CD, Dei Tos AP, Hohenberger P; EORTC Soft Tissue and Bone Sarcoma Group; PALETTE study group. Pazopanib for metastatic soft-tissue sarcoma (PALETTE): a randomised, double-blind, placebo-controlled phase 3 trial. Lancet. 2012 May 19;379(9829):1879-86. doi: 10.1016/S0140-6736(12)60651-5. Epub 2012 May 16. PMID 22595799
- [Background] Tap WD, Jones RL, Van Tine BA, Chmielowski B, Elias AD, Adkins D, Agulnik M, Cooney MM, Livingston MB, Pennock G, Hameed MR, Shah GD, Qin A, Shahir A, Cronier DM, Ilaria R Jr, Conti I, Cosaert J, Schwartz GK. Olaratumab and doxorubicin versus doxorubicin alone for treatment of soft-tissue sarcoma: an open-label phase 1b and randomised phase 2 trial. Lancet. 2016 Jul 30;388(10043):488-97. doi: 10.1016/S0140-6736(16)30587-6. Epub 2016 Jun 9. PMID 27291997
- [Background] Li J, Qin S, Xu J, Xiong J, Wu C, Bai Y, Liu W, Tong J, Liu Y, Xu R, Wang Z, Wang Q, Ouyang X, Yang Y, Ba Y, Liang J, Lin X, Luo D, Zheng R, Wang X, Sun G, Wang L, Zheng L, Guo H, Wu J, Xu N, Yang J, Zhang H, Cheng Y, Wang N, Chen L, Fan Z, Sun P, Yu H. Randomized, Double-Blind, Placebo-Controlled Phase III Trial of Apatinib in Patients With Chemotherapy-Refractory Advanced or Metastatic Adenocarcinoma of the Stomach or Gastroesophageal Junction. J Clin Oncol. 2016 May 1;34(13):1448-54. doi: 10.1200/JCO.2015.63.5995. Epub 2016 Feb 16. PMID 26884585
- [Background] Li J, Qin S, Xu J, Guo W, Xiong J, Bai Y, Sun G, Yang Y, Wang L, Xu N, Cheng Y, Wang Z, Zheng L, Tao M, Zhu X, Ji D, Liu X, Yu H. Apatinib for chemotherapy-refractory advanced metastatic gastric cancer: results from a randomized, placebo-controlled, parallel-arm, phase II trial. J Clin Oncol. 2013 Sep 10;31(26):3219-25. doi: 10.1200/JCO.2013.48.8585. Epub 2013 Aug 5. PMID 23918952
- [Background] Ding Q, Cheng X, Yang L, Zhang Q, Chen J, Li T, Shi H. PET/CT evaluation of response to chemotherapy in non-small cell lung cancer: PET response criteria in solid tumors (PERCIST) versus response evaluation criteria in solid tumors (RECIST). J Thorac Dis. 2014 Jun;6(6):677-83. doi: 10.3978/j.issn.2072-1439.2014.05.10. PMID 24976990
- [Background] Verger E, Salamero M, Conill C. Can Karnofsky performance status be transformed to the Eastern Cooperative Oncology Group scoring scale and vice versa? Eur J Cancer. 1992;28A(8-9):1328-30. doi: 10.1016/0959-8049(92)90510-9. PMID 1515244
- [Background] Li J, Zhao X, Chen L, Guo H, Lv F, Jia K, Yv K, Wang F, Li C, Qian J, Zheng C, Zuo Y. Safety and pharmacokinetics of novel selective vascular endothelial growth factor receptor-2 inhibitor YN968D1 in patients with advanced malignancies. BMC Cancer. 2010 Oct 5;10:529. doi: 10.1186/1471-2407-10-529. PMID 20923544
- [Background] Cirillo M, Venturini M, Ciccarelli L, Coati F, Bortolami O, Verlato G. Clinician versus nurse symptom reporting using the National Cancer Institute-Common Terminology Criteria for Adverse Events during chemotherapy: results of a comparison based on patient's self-reported questionnaire. Ann Oncol. 2009 Dec;20(12):1929-35. doi: 10.1093/annonc/mdp287. Epub 2009 Jul 17. PMID 19622510